CLINICAL TRIAL: NCT05994781
Title: A Prospective Researcher-led Clinical Study to Evaluate the Effectiveness and Safety of the Application of Neopep-S-based Easy Dew MD Regen Cream in Partial Layer Skin Transplantation
Brief Title: A Prospective Researcher-led Clinical Study of Neopep-S-based EasyDew MD Regen Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun-ji Kim (Industry)
Responsible Party: Sponsor-Investigator, Eun-ji Kim, Clinical Trial Manager, CGBio Inc.
Organization: CGBio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G2205
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment (No Intervention): The control group is a non-treatment group, and for 3 months after the procedure, general moisturizers that have been used or will be used are available.
- Treatment (Experimental): In the case of the study group among the subjects of the clinical study, The experimental group apply an appropriate amount of EasyDew MD Regen Cream twice a day (morning and evening) and can be absorbed well.
  Interventions: Device: EasyDew MD regen cram

INTERVENTIONS:
Device: EasyDew MD regen cram — No intervention
  Other Names: No treatment
  Arms: Treatment

SUMMARY:
This clinical study is conducted prospectively for 3 months after medical device treatment.

It is a comparative clinical study of the leading control group.

DETAILED DESCRIPTION:
Subjects need tissue transplantation to repair skin defects, so partial layer skin transplantation is performed. After proceeding, the patient is no longer subject to exudation. Subjects (and/or legal representatives) have agreed in writing to participate in the clinical study Perform a post-screening test.

Evaluating the screening test results, meeting the selection criteria, and meeting the exclusion criteria those who do not are registered for clinical research.

In the case of the study group among the subjects of the clinical study, whether partial layer skin transplantation was performed or not, Apply an appropriate amount of EasyDew MD Regen Cream twice a day (morning and evening) and can be absorbed well.

The control group is a non-treatment group, and for 3 months after the procedure. General moisturizers that have been used or will be used are available. The control group's Moisturizer is recommended twice a day (morning and evening) on whether skin grafts are collected or not Apply and allow good absorption. After applying medical devices and moisturizers for clinical research, the progress will be observed for 3 months, Subjects are a screening visit (Visit1), the day of medical device application (Visit2), and after medical device application.

Visit the research institution regularly for one month (Visit3) and three months after application (Visit4) for validity and it will be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 19
* Subjects with partial layer skin transplantation
* There is no evidence of infection in the skin transplant process, and exudate is no longer present a person who does not arise
* Decide to participate in this clinical study arbitrarily and in the written informed consent a person

Exclusion Criteria:

* showing signs of infection requiring antibiotic administration throughout the body or skin transplantation Case
* In situations where the requirements of a clinical study cannot be complied with
* When the researcher's judgment determines that the participation of the study is inappropriate (e.g. Kelloid personality)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
TEWL score | Before, after one month after application, 3 month after application
  Transepidermal water loss score/ No range of upper and lower score, the lower is best

SECONDARY OUTCOMES:
Investigator Global Assessment scale | Before, after one month after application, 3 month after application
  Assess the patient's overall condition /lowest 0 score ( best score) to highest 30 score( worst score)
Dermatology Life Quality Index | Before, after one month after application, 3 month after application
  Assess patient quality of life / lowest 0 score ( best score) to highest 4 score( worst score)
itching scale | Before, after one month after application, 3 month after application
  Evaluate the Itching scale / lowest 1 score ( best score) to highest 5 score( worst score)
VSS | Before, after one month after application, 3 month after application
  Vancouver Scar Scale/ No range of upper and lower score, the lower is best

CONTACTS AND LOCATIONS:
Overall Officials: Jihye Lee, Master, Study Director — CGBio Inc.
Locations (1):
- Ajou University Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No